CLINICAL TRIAL: NCT02748499
Title: Evaluation of the Healthy Beat Accupunch (HBA) Exercise Program for the Community Older Adults
Brief Title: Healthy Beat Accupunch (HBA) Exercise Program for Community Older Adults
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kaohsiung Medical University (Other)
Collaborators: National Science and Technology Council, Taiwan (Other Government)
Responsible Party: Principal Investigator, Kuei-Min Chen, Ph.D., RN., Professor, Kaohsiung Medical University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: KMUH-IRB-20140089-1
Record Dates: First submitted 2016-04-20; First posted 2016-04-22 (Estimated); Last update posted 2017-05-12 (Actual); Status verified 2017-05

CONDITIONS: Perceived Health Status; Sleep Quality
MeSH Terms: conditions — Sleep Initiation and Maintenance Disorders

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Healthy Beat Accupunch (Experimental): The HBA exercise program includes: 1) warm-up: 5 slow and gentle exercises to regulate qi, loosen up the body, and elevate the energy for a safe transition to the next phase, 2) accupunch: 14 low-to-medium speed exercises to punch the 14 meridians to enhance the cardiovascular-respiratory workout, and 3) relaxation: 5 low-speed, muscle relaxing exercises with deep breaths to sooth the body and mind. It is conducted 3 times per week and 40 minutes per practice.
  Interventions: Other: Healthy Beat Accupunch (HBA) exercise program
- Control (Active Comparator): The control group maintains daily activities.
  Interventions: Other: Control

INTERVENTIONS:
Other: Healthy Beat Accupunch (HBA) exercise program — HBA has three phases and takes 40 minutes to complete.
  Arms: Healthy Beat Accupunch
Other: Control — Participants maintain their daily acitvities.
  Arms: Control

SUMMARY:
This study aimed to test the effects of a 12-month Healthy Beat Accupunch (HBA) exercise program on the perceived health status and sleep quality of the community-dwelling older adults.

DETAILED DESCRIPTION:
Phase I: A cluster randomized controlled trial was used to test the effects of a six-month, instructor-led Healthy Beat Accupunch (HBA) exercise program on the perceived health status and sleep quality of the community-dwelling older adults. Through the use of convenience sampling strategy, eight community care centers with 232 older adults in Kaohsiung were recruited and randomly assigned based on their community care centers to a HBA experimental group or a wait-list control group. Participants in the experimental group received the HBA exercise program led by trained and certified instructors, three times per week, 40 minutes per practice for six months; participants in the wait-list control group continued with their regular daily activities. One pre-test and two post-tests, three months apart, were conducted. Phase II: Using the same method as in the phase I, participants from the phase I continued practicing the HBA exercise program, but guided by a DVD, for another six months. The feasibility, compliance, and effectiveness of the DVD-led HBA exercise program on the community-dwelling older adults were tested, and another two post-tests, three months apart, were conducted on the same outcome measurements as in the phase I.

ELIGIBILITY:
Inclusion Criteria:

* community-dwelling older adults aged 65 and over
* Mandarin or Taiwanese speakers
* able to stand and walk without assistive devices
* cognitive alert and able to verbally state their name, address, and answer questions

Exclusion Criteria:

* participants with severe and acute cardiovascular, musculoskeletal, or pulmonary illnesses

Ages: 65 Years to 100 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 232 (Actual)
Dates: Start 2014-07-12 (Actual); Primary Completion 2017-05-05 (Actual); Study Completion 2017-05-05 (Actual)

PRIMARY OUTCOMES:
Perceived health status measured by SF-12 Health Survey | 12 months
  measured by SF-12 Health Survey

SECONDARY OUTCOMES:
Sleep quality measured by Pittsburge Sleep Quality Index (PSQI) | 12 months
  measured by Pittsburge Sleep Quality Index (PSQI)

CONTACTS AND LOCATIONS:
Overall Officials: Kuei-Min Chen, Ph.D., Principal Investigator — Kaohsiung Medical University

IPD SHARING:
Plan to Share IPD: No